CLINICAL TRIAL: NCT03326999
Title: Evaluating the Addition of Obturator Nerve Block to Adductor Canal Block for Total Knee Arthroplasty
Brief Title: Does Adding an Additional Numbing Medication Injection in the Thigh Help With Pain Control After Knee Replacement Surgery?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Christina Jeng, Christina Jeng MD Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 17-2153
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Results first posted 2020-08-26 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Knee Osteoarthritis; Knee Rheumatism
Keywords: adductor canal regional block; obturator nerve regional block; total knee arthroplasty; knee replacement surgery; Knee rheumatoid arthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two arms: one arm will receive adductor canal block and obturator nerve block with the local anesthetic bupivacaine; second arm will receive adductor canal block with bupivacaine and obturator nerve block with saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational arm (Experimental): Patients in this arm will receive adductor canal regional block with bupivacaine and obturator nerve regional block with bupivacaine
  Interventions: Drug: Obturator nerve regional block; Drug: Adductor canal regional block
- Control arm (Sham Comparator): Patients in this arm will receive adductor canal regional block with bupivacaine and obturator nerve regional block with saline
  Interventions: Drug: Adductor canal regional block; Drug: Saline

INTERVENTIONS:
Drug: Obturator nerve regional block — Obturator nerve regional block involves the injection of a local anesthetic called bupivacaine into the upper thigh.
  Other Names: bupivacaine
  Arms: Investigational arm
Drug: Adductor canal regional block — Adductor canal regional block, which involves injecting numbing medication in the thigh region for pain control.
Drug: Saline — Saline as placebo comparator
  Arms: Control arm

SUMMARY:
One common anesthetic that is performed for total knee replacement surgery is spinal anesthesia with an adductor canal regional block, which involves injecting numbing medication in the thigh region for pain control after surgery. The aim of this study is to determine whether the addition of another regional block called obturator nerve block, which involves injecting numbing medication in the upper thigh region, will improve pain control after surgery while not sacrificing mobility after surgery.

DETAILED DESCRIPTION:
There is currently no consensus on the optimal strategy that provides the most effective postoperative analgesia while preserving ambulation and limiting side effects such as nausea and vomiting. The clinical team's hypothesis is that the obturator nerve block in addition to adductor canal block can target both the anterior and posterior distribution of nerves to the knee to provide superior analgesia while not limiting ambulation. To test this hypothesis, the clinical team will compare the rate of IV opioid consumption in patients who receive a combination of adductor canal block and obturator nerve block at the surgical site versus patients who receive adductor canal block alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo total knee arthroplasty
* Planned use of regional anesthesia for procedure
* Willing and able to provide informed consent

Exclusion Criteria:

* Patients on immunosuppressive therapy
* Patients with history of diabetes
* Patients with lower limb neuropathy
* Patients with history of chronic opioid use for > 3 months, including but not limited to, fentanyl, morphine, oxycodone, methadone
* Patients with known allergy or intolerance to any drug used in the study
* Patients with history of alcohol or drug abuse
* Patients with history of intolerance of nonsteroidal anti-inflammatory drugs
* Patients with hepatic or renal insufficiency
* ASA score of 4 or greater

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Jeng, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Runge C, Borglum J, Jensen JM, Kobborg T, Pedersen A, Sandberg J, Mikkelsen LR, Vase M, Bendtsen TF. The Analgesic Effect of Obturator Nerve Block Added to a Femoral Triangle Block After Total Knee Arthroplasty: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):445-51. doi: 10.1097/AAP.0000000000000406. PMID 27171822

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in October with enrollment from December 2017 through December 2018.
Groups:
- Investigational Arm: Patients in this arm received adductor canal regional block with bupivacaine and obturator nerve regional block with bupivacaine
- Control Arm: Patients in this arm received adductor canal regional block with bupivacaine and obturator nerve regional block with saline
Period: Overall Study
Arm/Group | Investigational Arm | Control Arm
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bupivacaine Arm: Patients in this arm received adductor canal regional block with bupivacaine and obturator nerve regional block with bupivacaine
- Saline Control Arm: Patients in this arm received adductor canal regional block with bupivacaine and obturator nerve regional block with saline
- Total: Total of all reporting groups
Arm/Group | Bupivacaine Arm | Saline Control Arm | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (7.5) | 66.7 (7.3) | 67.3 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 13 | 12 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 18 | 18 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 5 | 13
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.72 (4.85) | 28.65 (5.05) | 29.68 (5.02)

OUTCOME MEASURES:

1. Primary Outcome: Morphine Equivalence Consumption
Description: Total amount of opioids consumed
Time Frame: up to 24 hours after surgery
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Bupivacaine Arm | Saline Control Arm
Number analyzed (Participants) | 30 | 30
MME | 12.6 (6.37) | 18.85 (7.74)

2. Secondary Outcome: Pain Score
Description: Likert scale ranging from 0-10 - 0 being no pain, and 10 being the worst pain ever experienced
Time Frame: 1, 6, 12, and 24 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine Arm | Saline Control Arm
Number analyzed (Participants) | 30 | 30
score on a scale
  1 hour | 0.17 (0.64) | 0.23 (1.28)
  6 hours | 2.27 (2.82) | 2.77 (2.71)
  12 hours | 4.10 (2.92) | 5.13 (2.22)
  24 hours | 6.10 (2.66) | 7.00 (2.24)

3. Secondary Outcome: Number of Participants With Nausea or Vomiting
Description: Yes or No responses when the subject is asked if the subject is feeling nauseous or has vomited
Time Frame: up to 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine Arm | Saline Control Arm
Number analyzed (Participants) | 30 | 30
Participants | 11 | 16

4. Secondary Outcome: Time to Ambulation
Description: The length of time that it takes before the patient is first able to walk with assistance after surgery as assessed by a physical therapist.
Time Frame: on postoperative day 1 after surgery
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Bupivacaine Arm | Saline Control Arm
Number analyzed (Participants) | 30 | 30
hours | 8.98 (8.13) | 7.87 (8.49)

5. Secondary Outcome: Time to Breakthrough Pain Medication
Description: Time before pain medication needed for breakthrough pain
Time Frame: up to post operative day 2 after surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Bupivacaine Arm | Saline Control Arm
Number analyzed (Participants) | 30 | 30
minutes | 872.54 (1044.07) | 510.13 (420.69)

6. Secondary Outcome: Analgesia Satisfaction Score
Description: Analgesia Satisfaction Score - Full scale from 0-10 with higher score indicating higher satisfaction.
Time Frame: 2 weeks after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine Arm | Saline Control Arm
Number analyzed (Participants) | 30 | 30
score on a scale | 9.24 (0.93) | 8.59 (2.08)

ADVERSE EVENTS:
Time Frame: 2 weeks post surgery
Arm/Group | Investigational Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT03326999/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT03326999/SAP_001.pdf